CLINICAL TRIAL: NCT02580656
Title: An Open Trial of Metacognitive Therapy for Anxiety and Depression in Cancer (OMAC Study)
Brief Title: An Open Trial of Metacognitive Therapy for Anxiety and Depression in Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Peter Fisher, Dr, University of Liverpool
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UoL001166
Record Dates: First submitted 2015-09-27; First posted 2015-10-20 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Anxiety; Depression; Cancer
MeSH Terms: conditions — Anxiety Disorders; Depression; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metacognitive Therapy (Experimental): Metacognitive Therapy (MCT) is a brief psychological intervention which will be delivered over a course of six, one hour weekly sessions. Treatment will follow a manualised protocol.
  Interventions: Behavioral: Metacognitive Therapy

INTERVENTIONS:
Behavioral: Metacognitive Therapy — MCT helps patients to understand the deleterious and counterproductive effects of responding to negative thoughts and feelings with worry and rumination. Treatment aims to enable patients to exert greater metacognitive control over their worry and rumination. The positive and negative metacognitive beliefs that keep perseverative thinking in place are modified, using verbal and behavioural reattribution and through specifically designed therapeutic methods.
  Other Names: MCT

SUMMARY:
Survival rates in cancer continue to improve, with over 2 million adult cancer survivors in the United Kingdom, projected to increase to 4 million by 2030. Around 25% of these survivors require treatment for clinical levels of emotional distress. The investigators will conduct a phase I open trial to test the potential efficacy of MCT in cancer survivors.

DETAILED DESCRIPTION:
Survival rates in cancer continue to improve, with over 2 million adult cancer survivors in the United Kingdom, projected to increase to 4 million by 2030. Around 25% of these survivors require treatment for clinical levels of emotional distress. There is scope for improvements in the efficacy of current pharmacological and psychological interventions. Reflecting this limited efficacy in the face of the need for psychological treatment, the National Cancer Survivorship Research Initiative highlighted development and evaluation of practically feasible interventions for depression and anxiety in cancer survivors as an urgent research priority. It is recognised that current influential psychotherapeutic approaches need to be modified to meet the specific needs associated with cancer. However modifications have been pragmatic rather than theory-driven and have not improved efficacy.

This study addresses the stages of 'development' and 'piloting and feasibility' in intervention development, albeit with a relatively well-defined starting point given existing evidence for efficacy of MCT in other settings and promising preliminary evidence of applicability in cancer. The investigators will conduct a phase I open trial to test the potential efficacy of MCT in cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Cancer diagnosis at least 6 months previously
* Scoring >15 on the Hospital Anxiety and Depression Scale Total
* Stable on, or free from, psychotropic medication

Exclusion Criteria:

* History of psychotic disorder, learning disability, or organic mental disorder
* Risk of self-harm or suicide warranting immediate intervention
* In palliative phase of treatment
* Being considered for risk-reducing or reconstructive surgery within 1 year
* Concurrent psychological treatment
* Cognitive impairment precluding informed consent or participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-01; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS-Total) | Change in HADS total following the course of the six week intervention and over the six month follow-up
  A general measure of anxiety and depression used in people

CONTACTS AND LOCATIONS:
Overall Officials: Peter FISHER, PhD, Principal Investigator — University of Liverpool
Locations (1):
- Royal Liverpool and Broadgreen NHS Trust, Liverpool, Merseyside, United Kingdom